CLINICAL TRIAL: NCT01268761
Title: Usefulness of GnRH Antagonist Administration in the Treatment of Early Ovarian Hyperstimulation Syndrome
Brief Title: GnRH Antagonist for Treatment of Early Ovarian Hyperstimulation Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Juan Giles, Principal Investigator; Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0810-C-052-JG
Record Dates: First submitted 2010-12-23; First posted 2010-12-31 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Ovarian Hyperstimulation Syndrome; Effects of Gonadotropin; Oocyte Maturation
Keywords: Ovarian hyperstimulation syndrome (OHSS); GnRH antagonist; Ascitis.
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — cetrorelix; Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRH antagonist (Experimental): • GnRH antagonist (Cetrorelix 0.25)
  Interventions: Drug: GnRH antagonist (Cetrorelix)
- Placebo (saline solution) (Placebo Comparator): • Placebo (saline solution)
  Interventions: Drug: Placebo (saline solution)

INTERVENTIONS:
Drug: GnRH antagonist (Cetrorelix) — •GnRH antagonist (Cetrorelix 0.25) during 7 days beginning administration the second day of oocyte retrieval
  Arms: GnRH antagonist
Drug: Placebo (saline solution) — • Placebo (saline solution) 1 ampoule every 24 hours during 7 days beginning administration the second day of oocyte retrieval
  Arms: Placebo (saline solution)

SUMMARY:
The aim of this study is to analyze the effectiveness of GnRh antagonist in the treatment of early ovarian hyperstimulation syndrome.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome (OHSS) is a serious complication of ovarian stimulation protocols. Gonadotrophin-releasing hormone (GnRH) antagonist administration in the luteal phase was recently proposed as a new approach for the management of patients with established severe OHSS We analyze the response of egg donors with moderate- severe early ovarian hyperstimulation syndrome after a GnRH antagonist stimulation protocol to the administration of a daily doses of GnRH antagonist (Cetrorelix 0.25) during 7 days after the second day of oocyte retrieval compared with placebo (saline solution).

ELIGIBILITY:
Inclusion Criteria:

* Egg donors
* Volunteers.
* 18-35 years old
* Healthy
* BMI < 30
* OHHS after oocyte retrieval defined as ascitis > 9 cm2 associate to abdominal pain, sickness, abdominal distention,or haematocrit (Ht) >45% an white blood cell count >15,000/mm3 or creatine > 1.2 mg/dl or transaminases > 40 IU/liter

Exclusion Criteria:

* BMI > 30
* Allergy to GnRH antagonist

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ultrasound | one week
  Ultrasound measurements: ascitis and ovarian size
Blood measurements | one week
  Blood measurements: hyperstimulation biomarkers, liver and kidney function and hormonal profile.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Giles, MD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain